CLINICAL TRIAL: NCT00203151
Title: A Multi-National, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Parallel Group Study to Assess the Efficacy, Tolerability and Safety of Edratide for Subcutaneous Injection in Systemic Lupus Erythematosus (SLE)
Brief Title: A Study to Evaluate the Tolerability, Safety and Effectiveness of Edratide in the Treatment of Lupus
Acronym: PRELUDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: TV-4710/201 did not meet its primary endpoints in patients with SLE
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Rivka Kreitman, Ph.D., Vice President, Innovative Research & Development, Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV-4710/201
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — edratide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: edratide
- 2 (Placebo Comparator)
  Interventions: Drug: edratide

INTERVENTIONS:
Drug: edratide — 0.5 mg, 1.0 mg, 2.5 mg injection once weekly

SUMMARY:
It is thought that Edratide may be able to reduce the symptoms of SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent
2. Between the ages of 18 and 65 years (inclusive)
3. Fulfilled at least 4 ACR classification criteria
4. SLE patients with moderate, active disease
5. Subjects on stable dose of SLE medications for at least 4 weeks before randomization.
6. Women of child-bearing potential must practice a medically acceptable method of contraception..
7. Must understand the requirements of the study and agree to comply with the study protocol.

Exclusion Criteria:

1. Any condition which the investigator feels may interfere with participation in the study.
2. Subjects having a history of chronic infection
3. Subjects with a history of immunodeficiency syndrome or malignancy,
4. Subjects who received any investigational medication (including DHEA) within 3 months prior to randomization,
5. Subjects treated with any cytotoxic agents in the 3 months prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2005-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Improvement of Disease Activity Score | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Goldsatub, Ph.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.

REFERENCES:
- [Derived] Urowitz MB, Isenberg DA, Wallace DJ. Safety and efficacy of hCDR1 (Edratide) in patients with active systemic lupus erythematosus: results of phase II study. Lupus Sci Med. 2015 Aug 11;2(1):e000104. doi: 10.1136/lupus-2015-000104. eCollection 2015. PMID 26301100